CLINICAL TRIAL: NCT05470335
Title: Patient Comfort, Success Rate, Procedure Time and Complications During Sheath Insertion by Nurses and Physicians in Connection With Invasive Examination and Treatment of Cardiac Patients
Brief Title: Nurse-led Sheath Insertion in Cardiac Patients
Acronym: NUSHI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zealand University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMN-2021-08143
Record Dates: First submitted 2022-05-31; First posted 2022-07-22 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- physician insertion (No Intervention): radial sheath insertion is performed by physicians
- nurse insertion (Experimental): radial sheath insertion is performed by nurses
  Interventions: Procedure: nurse-led sheath insertion

INTERVENTIONS:
Procedure: nurse-led sheath insertion — radial sheaths for coronary examination and intervention are performed by experienced nurses
  Arms: nurse insertion

SUMMARY:
The aim of project NUSHI is to elucidate, that radial sheath insertion can be performed by nurses and physicians with the same level of comfort and safety.

DETAILED DESCRIPTION:
Background: Insertion of sheath in the radial artery in connection with examination and treatment of patients with coronary artery disease is usually performed by specialized invasive cardiologists or trainees. Whether sheath insertion can be performed by nurses with the same level of comfort and pain is uncertain.

Eligibility: Patients referred for coronary angiography (CAG) and/or percutaneous coronary intervention (PCI) due to suspicion of coronary artery disease are included

Randomization: Patients are randomized 1:1 to sheath insertion by nurse or physician

Methods: Insertion of 5 or 6 radial sheaths is performed in local anesthesia

Outcome measures: Comfort and pain level is registered from immediately after sheath insertion until start of CAG/PCI.

Additional outcome measures: Oximetry test is performed immediately after sheath removal - and repeated after 1 month in case of occlusion. Any complication is recorded from the patient enters the wake-up room until discharge.

All patients are contacted after 1 year in order to register adverse events.

ELIGIBILITY:
Inclusion Criteria:

* patients suspected of having coronary artery disease
* with normal puls oxymetry on the right hand
* understands patient information and accepts to participate

Exclusion Criteria:

* under consideration for cardiac valve replacement
* systolic blood pressure persistently >180 mmHg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
pain level | through study completion, an average of 1 year
  pain level during sheath insertion is measured using a 1 to 10 point numeric rating scale. For pain registration: 0 is no pain and 10 the worst imaginable pain.
comfort level | through study completion, an average of 1 year
  comfort level during sheath insertion is measured using a 1 to 10 point numeric rating scale. For comfort: 0 is no comfort at all and 10 is the best imaginable comfort.

SECONDARY OUTCOMES:
success rate | through study completion, an average of 1 year
  success rate with regard to successful sheath insertion is assured
time consumption | through study completion, an average of 1 year
  time consumption for both groups
convertion | through study completion, an average of 1 year
  successful conversion yes/no from physician to nurse or from nurse to physician determined by the possibility to accomplish the diagnostic or therapeutic procedure
complications | through study completion, an average of 1 year
  occurrence of radial occlusion, perforation, pseudoaneurysm, and compartment syndrome

CONTACTS AND LOCATIONS:
Overall Officials: Henning Kelbæk, MD, Principal Investigator — Chief Physician
Locations (1):
- Zealand University Hospital, Roskilde, Danmark, Denmark

IPD SHARING:
Plan to Share IPD: No